CLINICAL TRIAL: NCT05151549
Title: A Prospective Evaluation of Carilizumab Combined With Concurrent Chemoradiotherapy in High-risk PD-L1 Positive Stage III-IVA Cervical Cancer One-arm Phase II Clinical Study
Brief Title: A Study of Carilizumab Combined With Concurrent Chemoradiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCHIIT103
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer
Keywords: immunotherapy; PD-1 checkpoint inhibitor; concurrent chemoradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in this study.Participants will be given intravenous administration of Camrelizumab (200mg) ,Cisplatin(40mg/m²) or Carboplatin(AUC 2) and Radiotherapy. After completing 17 cycles of concurrent chemoradiation, the Participants will continue to use camrelizumab as maintenance therapy until one year.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab , Cisplatin or Carboplatin (Experimental): Participants will be given intravenous administration of Camrelizumab (200mg) ,Cisplatin(40mg/m²) or Carboplatin(AUC 2) and Radiotherapy. After completing 17 cycles of concurrent chemoradiation, the Participants will continue to use camrelizumab as maintenance therapy until one year.
  Interventions: Drug: Camrelizumab; Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Drug: Camrelizumab — 200mg/3weeks
Drug: Cisplatin or Carboplatin — Cisplatin (40mg/m²), every week Carboplatin(AUC 2)

SUMMARY:
This is a one-arm phase II clinical study. In patients with stage III-IVA cervical cancer with pelvic lymph nodes > 2cm, positive para-aortic lymph nodes, or lymph node metastases > 2, patients with positive PD-L1 expression (CPS score ≥1) were treated with cararizumab combined with conventional concurrent chemoradiotherapy and immunomaintenance therapy for one year. To evaluate the efficacy and safety of carilizumab in combination with concurrent chemoradiotherapy and subsequent maintenance therapy.

DETAILED DESCRIPTION:
The patient received neoadjuvant therapy once every three weeks for a total of seventeen cycles. From the first day of treatment, the patient will undergo concurrent chemoradiation for 5 weeks.The chemotherapy drug is cisplatin or carboplatin every week for 5 weeks. After the end of concurrent chemoradiation, the patient will continue to use camrelizumab as maintenance therapy until one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Understand the research procedures and content, and voluntarily sign informed consent
3. Histologically or cytologically confirmed squamous cell carcinoma, adenocarcinoma, or stage III-IVA cervical carcinoma with adenocarcinoma;
4. According to RECIST 1.1 criteria, subjects must have at least one of the following risk factors demonstrated by CT or MRI or PET-CT:1) Pelvic lymph nodes with short diameter ≥20mm and para-arterial lymph nodes with short diameter ≥10mm;2)The number of lymph nodes > 2 (single lymph node with short diameter ≥10mm);
5. CT, MRI, or PET-CT showed no distant metastasis;
6. Expected survival period ≥ 3 months
7. ECOG score: 0-1
8. Subject will provide sufficient formalin fixed paraffin embedded (FFPE) specimens or sections of tumor archived tissue or fresh tissue that meet the test criteria and will be willing to undergo tumor biopsy for PD-L1 if required. The archived tissue must be a representative tumor specimen from less than 3 years old, or a series of unstained sections (not less than 4) of FFPE tumor tissue from less than 6 months old, and the relevant pathological report of the above specimens must be provided. Fresh tissue samples can be obtained by surgical resection or biopsy. The methods of biopsy include but are not limited to core needle biopsy, endoscopic resection or clamp biopsy (ensure sufficient tumor cells > 100); Fine needle aspiration and liquid based cytology (TCT) samples are not accepted (i.e. samples that lack complete tissue structure and provide only cell suspension and/or cell smear); Demineralized specimens of bone metastases were not accepted. For patients with pD-L1 negative initial archived tumor tissue samples, biopsies may be performed at screening, subject to patient consent, to provide fresh tissue prepared wax blocks or slices for retesting for PD-L1 status.
9. Investigator-assessed suitability for concurrent chemoradiotherapy;
10. The values of laboratory tests performed for screening must meet the following criteria:

    Blood test 1) Hemoglobin (HGB) ≥90 g/L; 2) Absolute count of neutrophils (ANC) ≥1.5×109 /L; 3) Platelet (PLT) ≥100×109 /L; Biochemical examination 1) Total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome allowed ≤5×ULN); 2) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (if liver metastasis exists, ALT and AST≤5×ULN); 3) Serum creatinine (Cr) ≤1.5×ULN or endogenous creatinine clearance ≥50mL/min (Cockcroft Gault formula);
11. Thyroid function indicators: thyroid stimulating hormone (TSH) and free thyroid hormone (FT3/FT4) were in the normal range; If TSH is not in the normal range, FT3 and FT4 can be grouped if they are in the normal range.
12. The subjects can be followed up regularly, have good communication with the researchers, and complete the study in accordance with the provisions of the study.

Exclusion Criteria:

1. Histological examination results are small cell (neuroendocrine) cervical cancer and mucinous adenocarcinoma
2. CT, MRI or PET-CT examination shows diffuse pelvic metastasis
3. CT, MRI or PET-CT examination shows distant metastasis (excluding retroperitoneal lymph node metastasis)
4. A patient with a previous malignancy (other than cured basal cell carcinoma of the skin or squamous cell carcinoma) should not participate in the study unless she had a complete response for at least 5 years prior to enrollment and was not expected to require additional antitumor therapy during the study period;
5. Active central nervous system (CNS) metastases, including symptomatic brain metastases,meningeal metastases or spinal cord compression, etc.Asymptomatic brain metastases can be included in the group (no progression for at least 4 weeks after radiotherapy and/or no neurological symptoms or signs after surgical resection, no need for treatment with glucocorticoids, anticonvulsants or mannitol)
6. Systemic chemotherapy, targeted therapy, anti-tumor biological therapy (such as tumor vaccine, cytokine or growth factor, etc.) have been performed before the study drug
7. The effect of major surgery or severe trauma before study medication has been eliminated within 14 days(Those who have undergone local anesthesia or percutaneous needle biopsy within 7 days and have recovered can be included in the group)
8. Participants received systemic corticosteroids (prednisone>10mg/day or equivalent dose) or other immunosuppressive drugs within 14 days before the study medication
9. Have active, known history of autoimmune diseases, including but not limited to systemic lupus erythematosus (sle), psoriasis, rheumatoid arthritis, inflammatory bowel disease, hashimoto's thyroiditis, except: type I diabetes, only by hormone replacement therapy can control the hypothyroidism, no systemic treatment of skin diseases, such as vitiligo, and has celiac disease control;
10. Complications that require immunosuppressive drug therapy or systemic treatment at immunosuppressive doses (prednisone > 10mg/ day or equivalent dose of the same drug); In the absence of active autoimmune disease, inhaled or topical steroids and doses > 10mg/ day of prednisone or equivalent doses of similar drugs are permitted;
11. Uncontrolled hypertension (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg) or pulmonary hypertension or unstable angina; Myocardial infarction or bypass or stent surgery within 6 months before administration; A history of chronic heart failure that meets New York Heart Association (NYHA) criteria of grade 3-4; Valvular disease of clinical significance; Severe arrhythmias requiring treatment, including QTc interval ≥470 ms (as calculated by Fridericia formula); Left ventricular ejection fraction (LVEF) < 50%; Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months before administration;
12. Other serious medical diseases, including but not limited to: uncontrolled diabetes, active digestive ulcer, active bleeding, etc.;
13. Actively infected persons requiring systemic treatment;
14. Previously or currently infected with active TUBERCULOSIS;
15. Previous history of interstitial lung disease;
16. Symptomatic and uncontrollable serous effusion such as peritoneal, pleural, or pericardial effusion;
17. Human immunodeficiency virus antibody (HIV-AB) positive; Active syphilis infection; Hepatitis C antibody (HCV-AB) positive, and HEPATITIS C virus RNA quantitative > the upper limit of detection unit normal value; Hepatitis B virus surface antigen (HBsAg) positive, and hepatitis B virus detection value > the upper limit of normal value of the detection unit;
18. The adverse reactions caused by previous treatment have not recovered to level 1 or below (CTCAE5.0) (except for alopecia and level 2 neurotoxicity caused by chemotherapy drugs);
19. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies (or any other antibody acting on the T cell costimulation or checkpoint pathway);
20. Previous radiation therapy has been performed for the area to be irradiated;
21. Use of live or attenuated vaccine within 28 days prior to the study administration;
22. Use of any other study drug or research device within 30 days prior to the study medication;
23. Those with a history of drug abuse or drug abuse upon inquiry;
24. Previous clear history of neurological or mental disorders, such as epilepsy, dementia, poor compliance;
25. Breastfeeding women who do not agree to stop breastfeeding;
26. Known allergy to recombinant humanized PD-1 monoclonal antibody or any of its excipients; Known history of allergic disease or severe allergic constitution;
27. The investigator considers that it is not suitable to participate in this clinical investigator due to various other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | immediately after the concurrent chemoradiation
  Proportional patient proportion to survival and non-progressive in the second year. Use RECIST 1.1 evaluation criteria for evaluation and the unit is 'years'.

SECONDARY OUTCOMES:
duration of response (DOR) | 1 year
  t refers to the time from the first evaluation of the tumor as CR or PR to the first evaluation as PD (Progressive Disease) or death from any cause. Use RECIST 1.1 evaluation criteria for evaluation and the unit is 'years'.
Progression-free survival (PFS) | 1 year
  The time span from the beginning of treatment of the tumor to the appearance of secondary growth of the tumor. It means that the tumor has basically not progressed at this stage. Use RECIST 1.1 evaluation criteria for evaluation and the unit is 'years'.
overall survival (OS) | 1 year
  Time from receiving treatment to death (for any reason). Evaluation based on follow-up and the unit is 'years'.
Disease Control Rate (DCR) | 1 year
  The proportion of patients whose tumors have shrunk or stabilized for a certain period of time, including complete remission, partial remission and stable cases. Use RECIST 1.1 evaluation criteria for evaluation and the unit is '%'.

CONTACTS AND LOCATIONS:
Overall Officials: Ke-qiang zhang, Principal Investigator — Hunan Cancer Hospital

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published work